CLINICAL TRIAL: NCT06104761
Title: The Effect of Instrument- Assisted Soft Tissue Mobilization on Upper Crossed Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam omran Grase, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IASTM
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: Effect of instrument assisted sopf tissue mobilization on upper cross syndrome
Who Masked: Participant, Outcomes Assessor
Masking Description: Double ( participant , Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Release Group (Experimental): Release of tight muscles in upper crossed syndrome
  Interventions: Other: Release group; Other: strength exercises and stretching for upper crossed syndrome
- Control group (Other): strength exercises and stretching for upper crossed syndrome
  Interventions: Other: strength exercises and stretching for upper crossed syndrome

INTERVENTIONS:
Other: Release group — i will make release for these muscles ( upper trapizius , levator scapulae , strenomastoid ) in addition to sub occipital fascia , then I will apply conventional physical therapy in form of stretching exercises (Trapezius (upper fibers) muscle , Levator scapulae muscle , Pectoralis major and Sternocleidomastoid muscles) and strengthening exercises for these muscles (Deep neck flexors, Trapezius (middle and lower fibers), Rhomboids and Serratus anterior muscles).
  Arms: Release Group
Other: strength exercises and stretching for upper crossed syndrome — I will apply conventional physical therapy in form of stretching exercises (Trapezius (upper fibers) muscle , Levator scapulae muscle , Pectoralis major and Sternocleidomastoid muscles) and strengthening exercises for these muscles (Deep neck flexors, Trapezius (middle and lower fibers), Rhomboids and Serratus anterior muscles).

SUMMARY:
This study will be a randomized controlled trial conducted to investigate the effect of myofascial release with IASTM on pain intensity level, cervical ROM, chest expansion, craniovertebral angle and kyphotic angle in upper crossed syndrome patients. A sample size of 52 will be randomly allocated to two group ,(26 participants in each group), by using computer-generated random number list Control group will recieve conventional physical therapy in form of stretching and strengthening and experimental group will recieve firstly myofascial release with IASTM then applying the same conventional physical therapy of control group . Both groups will recieve 3 sessions per week for 4 weeks .

DETAILED DESCRIPTION:
Upper crossed syndrome is characterized by the altered activation of specific muscles and postural deviations of the head, neck, and shoulders. Alterations in muscle activation include tightness of suboccipital and short erector spinae muscles of the neck, levator scapulae (LS), and upper trapezius (UT) muscles on the dorsal side crossed by tightness of pectoralis major (PM) and minor, sternocleidomastoid (SCM), and scalene muscles on the ventral side, and weakness of deep neck flexors (DNF) on the ventral side crossed by weakness of rhomboids, serratus anterior (SA), and middle and lower trapezius (LT) muscles on the dorsal side .

Because of UCS described as muscle imbalance pattern which located within the cervical and thoracic spine region. These imbalances have been shown to produce elevation and forward movement of the shoulders, winging of the scapula, and a forward extension of the head. These changes lead to overstress of the cervical cranial junction and shoulders, which can cause neck and/or jaw pain, headaches, and shoulder problems .

In this syndrome, the increased activity of accessory muscles of respiration disturbs the breathing, and the temporomandibular joint (TMJ) may develop osteoarthritis, resulting in chronic neck pain .

For the available literature, with the lack of evidence supporting about the effects of using myofascial release with IASTM on UCS patients. So the aim of this study was to investigate the effect of myofascial release with IASTM on pain intensity level, cervical ROM, chest expansion, craniovertebral angle and kyphotic angle in UCS patients.

ELIGIBILITY:
Inclusion Criteria:

- 1-Age ranged from 18 to 45 years . 2- All participants had intensity of neck pain on VAS (4-8) (moderate cases) . 3 - All participants had mechanical neck pain and FHP (craniovertebral angle CVA < 49) CVA of < 49) ..

4- All participants had kyphosis angle ≥45°.

Exclusion Criteria:

* 1- Malignancy. 2- Fractures of the cervical spine. 3- Cervical radiculopathy or myelopathy. 4- Vascular syndromes such as vertebrobasilar insufficiency. 5- Rheumatoid arthritis. 6- Neck or upper back surgery. 7- Taking anticoagulants. 8- Local infection.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Cervical range of motion | up to 4 weeks
  The ROM of the cervical spine was measured using CROM device and CROM measurements had established validity which contains sagittal plane inclinometer, frontal plane inclinometer and transverse plane inclinometer Total active cervical flexion range in upright sitting , Total active cervical rotation ROM (right and left) in upright sitting , Total active cervical extension in upright sitting., Total active side pending ROM (right and left) in upright sitting .
Chest Expansion | up to 4 weeks
  Tape measurement to measure chest expansion For the upper thoracic excursion, the tape measure placed at the level of the fifth thoracic spinous process and the third intercostal space at the midclavicular line For the lower thoracic excursion, the tape measure placed at the level of the 10th thoracic spinous process and the tip of the xiphoid process .
Cranio verteberal angle | up to 4 weeks
  Digitized camera will be used it wiil be taken from lateral view photograph of the subject in his\her usual standing posture and taken again to minimize image distortion, and therapist placed a circular spirit level at the base of the camera to ensure that the camera is perpendicular to the horizontal level. Next, the tragus of the subject's ear will be marked and a plastic pointer will be attached to the skin overlying the C7 vertebra. Once the photograph is obtained, the therapist will use image to measure FHP, quantified by the cranio-vertbral angle (CVA) (the angle between the horizontal lines passing through C7and a line extending from the tragus of the ear to C7 notably). Lesser CVA indicates greater FHP
Thoracic Kyphosis | up to 4 weeks
  Flexicurve ruler will be used to measure kyphosis The subject will be instructed to stand up straight and as tall as possible, and the flexicurve ruler will be aligned to the anterior-posterior curves of the spine from C7 to T12. The ruler will then placed flat on paper and its outline will be traced. A straight line was then drawn from the ruler position of C7 to T12 that corresponded to the length of thoracic kyphosis (l) and will be measured in cm. The height of the thoracic kyphosis (h) in cm will be determined by drawing a perpendicular line from the highest point in the thoracic curve to the point at which it will intersect the straight line drawn from C7 to T12. The index of kyphosis was calculated by applying the formula: (h/l ) x 100.
pain Intenisty level | up to 4 weeks
  Numeric Pain Rating Scale (NPRS) will be used to measure pain intensity level To assess pain intensity it is the most widely used tool for estimating both severity of pain and to judge the extent of pain relief. Patient will asked to select a point on a line drawn between two ends to express how intense he/she perceives pain. It composed of 10 cm long, anchored by two verbal descriptors (i.e., "no pain" and "worst imaginable pain". Patients are asked to rate "current" pain intensity or pain intensity "in the last 24 hours"